CLINICAL TRIAL: NCT04798703
Title: Phase I Exploratory Study of ONCOFID-P-B™ (PACLITAXEL-HYALURONIC ACID) Administered for 12 Consecutive Weeks Followed by Maintenance Therapy in BCG Unresponsive/ Intolerant Patients With Bladder Carcinoma in Situ (CIS)
Brief Title: Study of ONCOFID-P-B™ (PACLITAXEL-HYALURONIC ACID)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R39-17-01
Record Dates: First submitted 2020-12-02; First posted 2021-03-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-12

CONDITIONS: Bladder Carcinoma in Situ (CIS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONCOFID-P-B™ (PACLITAXEL-HYALURONIC ACID) (Experimental)
  Interventions: Drug: ONCOFID-P-B™ (PACLITAXEL-HYALURONIC ACID)

INTERVENTIONS:
Drug: ONCOFID-P-B™ (PACLITAXEL-HYALURONIC ACID) — 12 weekly intravesical instillations of ONCOFID-P-B™ (intensive treatment phase) followed by maintenance phase of the study, during which ONCOFID-P-B™ is furtherly administered once a month for 12 months in patients who achieved a complete response (CR) after the 12 weekly instillations.

SUMMARY:
Phase I exploratory, open-label, single arm, multicenter study to assess safety, tolerability and antitumor activity of ONCOFID-P-B™ therapy in adult patients with histologically confirmed diagnosis of bladder carcinoma in situ (CIS), who were unresponsive or intolerant to Bacillus Calmette-Guérin (BCG)-therapy.

Patients are initially treated with 12 weekly intravesical instillations of ONCOFID-P-B™ (intensive treatment phase). Patients who achieve a complete response (CR) after the 12 weekly instillations entered the maintenance phase of the study, during which ONCOFID-P-B™ is furtherly administered once a month for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed CIS of the bladder. A portion of patients up to 30% could have concomitant Ta and/or T1 lesions.
* Complete resection of papillary lesions before entering the trial in patients with concomitant CIS and papillary tumors.
* Patients were to be unresponsive or intolerant to BCG, had to have refused radical cystectomy or were not clinically suitable for cystectomy. Patients unresponsive to BCG were defined as patients for whom further BCG would be unlikely to be of benefit. This included all patients treated with an adequate course of induction plus maintenance BCG who either had persistent disease or who relapsed within 6 months of their last BCG treatment.
* Age ≥18 yrs.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Female in non-reproductive years (defined as surgically sterile or one year postmenopausal). Female of childbearing potential had to agree to practice complete abstinence or to use an effective contraceptive method.
* Able and willing to comply with scheduled visits, therapy plans, and laboratory tests required in the protocol.
* Signed and dated Independent Ethics Committee (IEC)-approved Informed Consent.

Exclusion Criteria:

* Any of the following in the previous 6 months: myocardial infarction, uncontrolled cardiac arrhythmia, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart enrolled cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis.
* Known hypersensitivity to paclitaxel or any of its constituents.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to treatment start.
* Muscle-invasive disease T2-T4.
* Previous or concomitant cancer of the upper urinary tract or the prostatic urethra.
* Prior (within the previous 3 years) or concurrent malignancies at other sites, except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri.
* Last intravesical immunotherapy dose administration <8 weeks prior to study entry. Patients had to have documentation of persistent or recurrent disease.
* Previous intravesical chemotherapy < 28 days prior to study entry with the exception of patients who underwent transurethral resection (TUR) < 7 days.
* Bladder capacity lower than 150 ml.
* Presence of significant urologic disease interfering with intravesical therapy.
* Concurrent enrollment or participation in another therapeutic clinical trial within 4 weeks preceding treatment start.
* Patients with known active substances and/or alcohol abuse.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with study participation or interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patients inappropriate for entry into the study or, in the opinion of the Investigator and/or the Sponsor, could compromise protocol objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) will be coded using MedDRA and their severity graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. | Safety data will be evaluated in the treated patient population through study completition, an average of 15 months.
  Overall safety profile evaluated based on clinical safety parameters (i.e. hematology and blood chemistry, urinalysis, vital signs and adverse events).
Laboratory test values will be graded according to the NCI CTCAE scale, v 4.03. | Safety data will be evaluated in the treated patient population through study completition, an average of 15 months.
  For each laboratory test included in the NCI CTCAE system, the incidence of abnormalities will be evaluated by considering the worst occurrence for each patient throughout the whole treatment period.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) - End of intensive treatment phase, | CRR will be evaluated after intensive treatment phase, at 12 weeks.
  Calculated as the proportion of patients who achieved a complete response after 12 weekly instillations of ONCOFID-P-B™.
CRR - End of maintenance phase | CRR will be evaluated after the end of the entire treatment period (intensive and maintenance), at 15 months.
  Calculated as the proportion of patients who achieved a complete response after the end of the entire treatment period (intensive + maintenance).
CRR - At 6 months | CRR will be evaluated at 6 months since treatment start.
  Calculated as the proportion of patients who achieved a complete response after 6 months since treatment start.
Rate of Overall Complete Response - Duration of Response (DoR), defined as the time from when criteria for Complete Response were first met until the first documented occurrence of CIS relapse or progression was reported. | CR will be evaluated at any time during the study up to 12 months after the end of treatment period
  Calculated as the proportion of patients who achieved complete response at any time during the study.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (2):
  - Istituto Europeo di Oncologia, Milan, Mi
  - IRCCS Humanitas, Rozzano, MI
- Spain (3):
  - Parc de Recerca Biomèdica de, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid